CLINICAL TRIAL: NCT00380471
Title: Treatment and Complication of Bath PUVA in Vitiligo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: src-pts-968
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Vitiligo
Keywords: bath PUVA
MeSH Terms: conditions — Vitiligo

INTERVENTIONS:
Device: Bath PUVA

SUMMARY:
The purpose of this study is to determine whether bath PUVA are effective in treatment of vitiligo and what is the complication of bath PUVA in vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Vitiligo

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Study Completion 2006-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Parviz Toossi, M.D., Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Skin Research Center, Shaheed Beheshti Medical University, Tehran, Iran